CLINICAL TRIAL: NCT02962518
Title: PRESSURE: Prospektive, Randomisierte Und Kontrollierte Untersuchung Von Lokaler Druckapplikation im Rahmen Der Keloid-Therapie Der Ohrmuschel
Brief Title: Pressure Device in the Treatment of Ear Keloids
Acronym: PRESSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Hoffmann, Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 68/14
Record Dates: First submitted 2016-11-04; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Keloid Ear
Keywords: Pressure Device; Clip; Triamcinolone; Fillet Technique
MeSH Terms: interventions — Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Standard Treatment (Active Comparator): Patients undergo surgery using the "fillet technique" and intra-lesional injections of triamcinolone 10mg /ml every 4 to 6 weeks for 6 months.
  Interventions: Procedure: Fillet Technique; Drug: Triamcinolone
- B Pressure Device (Experimental): Patients undergo surgery using the "fillet technique" and intra-lesional injections of triamcinolone 10mg /ml every 4 to 6 weeks for 6 months and are additionally treated with a non-customized pressure device.
  Interventions: Device: Pressure Device; Procedure: Fillet Technique; Drug: Triamcinolone

INTERVENTIONS:
Device: Pressure Device — Patients undergo surgery using the "fillet technique" and intra-lesional injections of triamcinolone 10mg /ml every 4 to 6 weeks for 6 months and they are additionally treated with a non-customized Pressure Device. The standardized clips (K. Egner, Dental Technique, Neu-Ulm, Germany) used in our study is available in two different sizes for smaller or larger defects. According to the guidelines of the German Society of Dermatology, patients are advised to wear the clip at least 16 hours per day. Medically approved transparent acrylate is used so that change in skin color and therefore amount of pressure can be observed at all times. Allergic or toxic skin involvement can be visualized through the transparent surface. Adjusting of the clip is done with one or two screws.
  Arms: B Pressure Device
Procedure: Fillet Technique — Patients undergo surgery using the fillet technique. To prevent the remaining skin from further damage, the meticulous skin preparation is performed either using the microscope or magnifying glasses. The keloid is "peeled" out of the excessive skin pocket. If necessary skin trimming is performed and non-resorbable monofilament single sutures are placed.
Drug: Triamcinolone — All patients received intra-lesional injections of tiamcinolone 10mg/ml every 4 to 6 weeks for 6 months.
  Other Names: Volon A

SUMMARY:
Keloids are benign cutaneous lesions, arising from proliferating fibroblasts. Keloids of the ear may occur after helix piercings and are difficult to treat, since they tend to form recurrences. Guidelines suggest multimodal therapy, however, recurrence rates remain high and prospective randomized trials are still missing.

To unravel the most effective combination of therapeutic options for keloids of the ear, 20 patients will be enrolled in a prospective, randomized trial. Patients either undergo surgery using the "fillet technique" and intra-lesional injections of triamcinolone 10mg /ml every 4 to 6 weeks for 6 months, or they are additionally treated with a non-customized pressure device.

DETAILED DESCRIPTION:
The prospective randomized controlled trial will be conducted at the Department of Otorhinolaryngology, Head and Neck Surgery, University Medical Center Ulm, Germany. 20 patients will be enrolled in the study. Prior to inclusion, informed written consent is obtained from each patient. Patients with immunodeficiency are not included, as well as patients with an infectious disease or patients with a missing capacity for consent. All patients undergo surgery using the fillet technique. To prevent the remaining skin from further damage, the meticulous skin preparation is performed either using the microscope or magnifying glasses. The keloid is "peeled" out of the excessive skin pocket. If necessary skin trimming is performed and non-resorbable monofilament single sutures are placed. The first intracutaneous injection of triamcinolone 10mg/ml is given before wound dressing is placed. A blanching of the lesion marks the endpoint of injection. Cutaneous sutures are removed after approximately 7 days. Injection of triamcinolone is repeated every 4 to 6 weeks for a total of 6 months. When removing the sutures, patients are randomized using consecutive sampling. Patients in group A are treated according to the protocol outlined above, having steroid injections for 6 months after surgical removal of the keloid. Group B involves patients who are additionally treated with non-customized pressure devices. The standardized clips (K. Egner, Dental Technique, Neu-Ulm, Germany) used in our study are available in two different sizes for smaller or larger defects. According to the guidelines of the German Society of Dermatology, patients are advised to wear the clip at least 16 hours per day. Medically approved transparent acrylate is used so that change in skin color and therefore amount of pressure can be observed at all times. Allergic or toxic skin involvement can be visualized through the transparent surface. Adjusting of the clip is done with one or two screws.

ELIGIBILITY:
Inclusion Criteria:

* Keloids of the helical rim of the ear

Exclusion Criteria:

* immunodeficiency
* infectious disease
* missing capacity for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Recurrence | 12 months
  Keloid recurrence

SECONDARY OUTCOMES:
Aesthetic scar outcome after treatment | 12 months
  assessed by visual analog scale (VAS) scores
Patients satisfaction | 12 months
  assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Hoffmann, Prof. Dr., Study Chair — Department of Otorhinolaryngology, Head and Neck Surgery, University Medical Center Ulm, Germany
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery, University Medial Center Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No